CLINICAL TRIAL: NCT01038609
Title: A Randomized, Multicenter, Single-Blind Study Comparing Hydrocodone/Acetaminophen Extended Release 10/650, Morphine Extended Release, and Acetaminophen to Placebo in Subjects With Acute Pain Following Bunionectomy
Brief Title: Hydrocodone/Acetaminophen for Acute Pain Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M12-058
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Pain
Keywords: Postoperative Pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Hydrocodone; Acetaminophen; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release) plus 1 placebo capsule (for morphine extended release), administered once every 12 hours, and 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release), administered once every 6 hours (for a total of 8 doses).
  Interventions: Drug: Placebo
- Acetaminophen (Active Comparator): 1 dose of 1 placebo capsule (for morphine extended release) plus 1 acetaminophen tablet, administered once every 12 hours, and 1 dose of 1 acetaminophen tablet, administered once every 6 hours (for a total of 8 doses).
  Interventions: Drug: Acetaminophen
- Morphine Extended Release (Active Comparator): 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release) plus 1 morphine extended release capsule, administered once every 12 hours, and 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release), administered once every 6 hours (for a total of 8 doses).
  Interventions: Drug: Morphine Extended Release
- Morphine Extended Release / Acetaminophen (Active Comparator): 1 dose of 1 morphine extended release capsule plus 1 acetaminophen tablet, administered once every 12 hours, and 1 dose of 1 acetaminophen tablet, administered once every 6 hours (for a total of 8 doses).
  Interventions: Drug: Acetaminophen; Drug: Morphine Extended Release
- Hydrocodone/Acetaminophen Extended Release (Experimental): 1 dose of 1 hydrocodone/acetaminophen extended release tablet plus 1 placebo capsule (for morphine extended release), administered once every 12 hours, and 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release), administered once every 6 hours (for a total of 8 doses).
  Interventions: Drug: Hydrocodone/Acetaminophen Extended Release

INTERVENTIONS:
Drug: Hydrocodone/Acetaminophen Extended Release
  Other Names: ABT-712
  Arms: Hydrocodone/Acetaminophen Extended Release
Drug: Acetaminophen
  Other Names: Tylenol
  Arms: Acetaminophen; Morphine Extended Release / Acetaminophen
Drug: Morphine Extended Release
  Other Names: Kadian
  Arms: Morphine Extended Release; Morphine Extended Release / Acetaminophen
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study was to evaluate analgesic efficacy and safety of hydrocodone/acetaminophen extended release compared to placebo in moderate to severe pain following primary unilateral first metatarsal bunionectomy.

DETAILED DESCRIPTION:
The bunionectomy was performed under regional anesthesia and propofol sedation. Perioperative anesthesia was standardized for all participants. Upon completion of surgery, designated study personnel ensured continued eligibility per the selection criteria of the protocol.

After an appropriate period of time following bunionectomy, participants who had a pain intensity score of ≥ 40 mm on a 100 mm visual analog scale (VAS) and moderate or severe pain intensity per the categorical pain intensity scale were eligible for randomization, in equal numbers, into 1 of 5 treatment arms. In order to maintain the single-blind nature of the study, all participants were dosed with study drug (active and/or placebo) every 6 hours.

ELIGIBILITY:
Inclusion Criteria:

- Subjects who were in general good health, experiencing moderate to severe pain following bunionectomy surgery and who were willing to remain confined for approximately 4 days following surgery for study procedures.

Exclusion Criteria:

* Subjects who underwent Base wedge osteotomy and/or Long-Z hart bunionectomy procedures
* Allergic reaction to study medications
* Pregnant or breastfeeding females
* Clinically significant lab abnormalities at screening
* Positive hepatitis testing at screening
* Clinically significant or uncontrolled medical disorders or illness at screening
* Active malignancy or chemotherapy
* Any history of drug or alcohol abuse/addiction
* Known or suspected history of human immunodeficiency virus (HIV); requires treatment with monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs) or butyrophenones
* History of major depressive episode or major psychiatric disorder
* Current systemic corticosteroid therapy
* Inability to refrain from smoking during or alcohol during stay at investigative site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Quintana Diez, MD, Study Director — AbbVie
Locations (4):
- United States (4):
  - Site Reference ID/Investigator# 26223, Peoria, Arizona
  - Site Reference ID/Investigator# 26302, Austin, Texas
  - Site Reference ID/Investigator# 26303, San Marcos, Texas
  - Site Reference ID/Investigator# 26304, West Jordan, Utah

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Started | 50 | 52 | 49 | 48 | 51
Completed | 49 | 51 | 48 | 47 | 50
Not Completed | 1 | 1 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Dosing Error | 0 | 0 | 0 | 1 | 1
Not completed — Death in the Family | 1 | 0 | 0 | 0 | 0
Not completed — Refusal of Blood Draws | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo | Total
Number analyzed (Participants) | 50 | 52 | 49 | 48 | 51 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (13.83) | 44.0 (12.93) | 40.2 (11.31) | 40.4 (13.16) | 45.2 (12.47) | 43.0 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 39 | 41 | 45 | 214
  Male | 5 | 8 | 10 | 7 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) Using the Pain Intensity Visual Analogue Scale (VAS)
Description: Participants assessed pain intensity on a 100 mm visual analogue scale (VAS) with 0 meaning "no pain" and 100 meaning the "worst pain imaginable". The SPID VAS score for 0 to 48 hours following initial study drug dose measured the cumulative pain intensity difference during treatment with higher mean SPID VAS scores indicating greater improvement from Baseline. The SPID score is a measure of the cumulative pain intensity difference during treatment and the area under the curve was estimated using the linear trapezoidal rule.
Time Frame: From time of first study drug administration to 48 hours following first study drug administration
Population: All randomized participants who received at least 1 dose of study drug. Analyses were performed based on the treatment participants actually received (as-treated).
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 50 | 52 | 49 | 48 | 51
scores on a scale | 720.5 (154.89) | 239.9 (151.41) | 614.4 (156.92) | 450.8 (159.62) | -57.6 (153.99)

2. Secondary Outcome: TOTPAR (Total Pain Relief)
Description: TOTPAR was the time-interval weighted sum of pain relief. Pain relief was assessed by participants' responses to how their pain relief was compared with the pain they had just before receiving the first dose of study drug: no relief, a little relief, some relief, a lot of relief, or complete relief. Higher mean TOTPAR scores indicate better pain relief. The TOTPAR score is a measure of the cumulative pain intensity difference during treatment and the area under the curve was estimated using the linear trapezoidal rule.
Time Frame: From time of first study drug administration to 48 hours following first study drug administration
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 50 | 52 | 49 | 48 | 51
scores on a scale | 65.9 (7.17) | 42.7 (7.01) | 49.5 (7.24) | 56.3 (7.34) | 32.9 (7.12)

3. Secondary Outcome: Participant's Global Assessment of Study Drug
Description: The participant's overall impression of the study drug was obtained on a 5-point categorical scale: excellent; very good; good; fair; poor.
Time Frame: From time of first study drug administration to 48 hours following first study drug administration
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 50 | 52 | 49 | 48 | 51
participants
  Excellent | 9 | 8 | 4 | 7 | 3
  Very Good | 15 | 16 | 19 | 20 | 17
  Good | 16 | 14 | 12 | 15 | 12
  Fair | 10 | 3 | 11 | 4 | 15
  Poor | 0 | 11 | 3 | 2 | 4

4. Secondary Outcome: Time to Perceptible and Meaningful Pain Relief
Description: The median time (minutes) from first perceptible pain relief (onset of pain relief) and time until first meaningful pain relief.
Time Frame: From time of first study drug administration to 12 hours following first study drug administration
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 50 | 52 | 49 | 48 | 51
minutes
  Time to Onset of Perceptible Pain Relief | 25.5 [17.0 to 30.0] | 32.0 [25.0 to 63.0] | 31.0 [22.0 to 44.0] | 22.5 [18.0 to 27.0] | 23.0 [16.0 to 37.0]
  Time to Onset of Meaningful Pain Relief | 62.5 [46.0 to 90.0] | 142.0 [76.0 to NA] — not available from Kaplan-Meier estimate | 101.0 [53.0 to NA] — not available from Kaplan-Meier estimate | 60.5 [49.0 to 83.0] | 220.0 [64.0 to NA] — not available from Kaplan-Meier estimate

5. Secondary Outcome: Participants With Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with treatment. If an adverse event meets any of the following criteria, it is considered a serious adverse event (SAE): results in death or is life-threatening, results in admission or prolongation of hospitalization, results in congenital anomaly or persistent or significant disability/incapacity, or is an important medical event requiring medical or surgical intervention to prevent serious outcome. AEs were categorized by severity (mild, moderate, severe) and relationship to treatment (probably, possibly, probably not, not related). Please see Adverse Events section below for more details.
Time Frame: AEs were recorded from study drug administration until 30 days following discontinuation of study drug (total 32 days); SAEs were recorded from the time informed consent was obtained until 30 days following discontinuation of study drug (total 51 days).
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 50 | 52 | 49 | 48 | 51
participants
  Any AE | 28 | 29 | 28 | 33 | 28
  Any AE at least "possibly" drug related | 23 | 23 | 23 | 24 | 19
  Any "severe" AE | 1 | 1 | 2 | 5 | 1
  Any SAE | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of study drug | 0 | 0 | 1 | 0 | 0
  Any AE leading to death | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Vital Signs Values Meeting Potentially Clinically Significant Criteria
Description: Potentially clinically significant criteria: Systolic blood pressure (BP) ≤90 mm Hg and ≥20 mm Hg decrease (low) or ≥180 mm Hg and ≥20 mm Hg increase (high); Diastolic BP ≤50 mm Hg and ≥15 mm Hg decrease (low) or ≥105 mm Hg and ≥15 mm Hg increase (high). Heart rate ≤50 beats per minute (bpm) and ≥15 bpm decrease (low) or ≥120 bpm and ≥15 bpm increase (high). Respiratory rate <10 respirations per minute (rpm) (low) or >24 rpm (high).
Time Frame: At specified intervals from Screening through 7 days after first dose of study drug
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 50 | 52 | 49 | 48 | 51
participants
  Systolic BP decrease | 3 | 6 | 8 | 2 | 5
  Systolic BP increase | 1 | 0 | 0 | 0 | 1
  Diastolic BP decrease | 2 | 5 | 6 | 5 | 2
  Diastolic BP increase | 0 | 0 | 2 | 0 | 0
  Heart rate decrease | 3 | 1 | 0 | 2 | 0
  Heart rate increase | 1 | 0 | 0 | 1 | 0
  Respiratory rate < 10 rpm | 0 | 0 | 0 | 0 | 0
  Respiratory rate > 24 rpm | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Chemistry Values Meeting Potentially Clinically Significant Criteria
Description: Potentially clinically significant criteria: alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≥3 times upper limit of normal (ULN); calcium ≤1.8 mmol/L.
Time Frame: At specified intervals from Screening through 7 days after first dose of study drug
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release / Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 50 | 52 | 49 | 48 | 51
participants
  ALT >= 3 * ULN | 1 | 2 | 3 | 0 | 0
  AST >= 3 * ULN | 1 | 2 | 3 | 0 | 0
  Calcium <= 1.8 mmol/L | 0 | 0 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: AEs were recorded from study drug administration until 30 days following discontinuation of study drug (total 32 days); SAEs were recorded from the time informed consent was obtained until 30 days following discontinuation of study drug (total 51 days).
Groups:
- Morphine Extended Release: 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release) and 1 morphine extended release capsule, administered once every 12 hours, and 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release), administered once every 6 hours (for a total of 8 doses).
- Morphine Extended Release/Acetaminophen: 1 dose of 1 morphine extended release capsule and 1 acetaminophen tablet, administered once every 12 hours, and 1 dose of 1 acetaminophen tablet, administered once every 6 hours (for a total of 8 doses).
- Hydrocodone/Acetaminophen Extended Release: 1 dose of 1 hydrocodone/acetaminophen extended release tablet and 1 placebo capsule (for morphine extended release), administered once every 12 hours, and 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release), administered once every 6 hours (for a total of 8 doses).
- Placebo: 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release) and 1 placebo capsule (for morphine extended release), administered once every 12 hours, and 1 dose of 1 placebo tablet (for hydrocodone/acetaminophen extended release), administered once every 6 hours (for a total of 8 doses).
Arm/Group | Acetaminophen | Morphine Extended Release | Morphine Extended Release/Acetaminophen | Hydrocodone/Acetaminophen Extended Release | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52 | 0/49 | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 19/50 | 21/52 | 26/49 | 27/48 | 20/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acetaminophen (N=50) | Morphine Extended Release (N=52) | Morphine Extended Release/Acetaminophen (N=49) | Hydrocodone/Acetaminophen Extended Release (N=48) | Placebo (N=51)
CONSTIPATION (Gastrointestinal disorders) | 0 | 3 | 1 | 3 | 3
DIARRHOEA (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 2
NAUSEA (Gastrointestinal disorders) | 6 | 7 | 11 | 16 | 9
VOMITING (Gastrointestinal disorders) | 1 | 4 | 6 | 7 | 3
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 1 | 2 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0
DIZZINESS (Nervous system disorders) | 4 | 4 | 9 | 6 | 3
HEADACHE (Nervous system disorders) | 6 | 8 | 9 | 8 | 5
SOMNOLENCE (Nervous system disorders) | 3 | 4 | 3 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.